CLINICAL TRIAL: NCT00146900
Title: Prevention of Post Traumatic Stress Disorder by Early Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Aria Shalev, Emeritus Professor of Psychiatry, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-27.06.03-HMO-CTIL; MH-
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Traumatic Events; Post-traumatic Stress Disorder; Treatment (psychological); Treatment (pharmacological); Prevention; SSRIs
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Escitalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Prolonged Exposure (CBT) (Experimental): Twelve 1.5 hours weekly sessions of Prolonged Exposure cognitive behavioral therapy
  Interventions: Procedure: Cognitive Behavioral Therapy
- Cognitive Therapy (Active Comparator): Twelve 1.5 hours weekly sessions of Cognitive Therapy without exposure to traumatic reminders.
  Interventions: Procedure: Cognitive Therapy
- SSRI (escitalopram) (Experimental): Twenty milligrams daily of escitalopram (blinded capsules)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Two concealed placebo pills resembling 10mg escitalopram tablets
  Interventions: Other: Placebo
- Waiting List (No Intervention): Twelve weeks of waiting list no intervention group

INTERVENTIONS:
Procedure: Cognitive Behavioral Therapy — 12 weekly 1.5 hours weekly session of cognitive behavioral therapy (Prolonged Exposure)
  Arms: Prolonged Exposure (CBT)
Procedure: Cognitive Therapy — 12 weekly 1.5 hours weekly session of cognitive therapy without exposure
  Arms: Cognitive Therapy
Drug: Escitalopram — Twelve weeks of treatment with Escitalopram at Max. daily dose of 20mg
  Other Names: SSRI
  Arms: SSRI (escitalopram)
Other: Placebo — Twelve weeks of treatment with placebo pills resembling the original Escitalopram 10mg tablets but containing no active substance
  Arms: Placebo

SUMMARY:
To prospectively evaluate the effect of early treatment (cognitive therapy (CT), cognitive-behavioral therapy (CBT) and escitalopram (SSRI) in preventing the occurrence of post-traumatic stress disorder in recent survivors of traumatic events.

DETAILED DESCRIPTION:
Consecutive civilian trauma survivors will be contacted, by phone, within five days of admission to Hadassah University Hospital in Jerusalem and asked about their early psychological responses to the event. A short telephone interview will be administered to consenting subjects, to evaluate the presence of acute stress disorder (ASD). Subjects with ASD (full or partial) and those who so desire will be invited to clinical assessment, which will take place within the next two weeks. Survivors with significant symptoms of post-traumatic stress disorder will be randomized to five arms of twelve-week long treatment: CBT, CT, SSRI/placebo and waiting list (WL) and start treatment immediately. Subjects will be allowed to decline one form of therapy. WL subjects will start therapy 12 weeks later. All subjects who had clinical interview will be interviewed again at four and seven months - and 14 months following trauma (phone interview).

ELIGIBILITY:
Inclusion Criteria:

* Adults survivors of traumatic events

Exclusion Criteria:

* Traumatic brain injury
* Lifetime psychosis
* Life time (prior) PTSD
* Medical conditions forbidding SSRIs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder (chronic) by CAPS scores. | Four months, seven months, 14 moths, two years

SECONDARY OUTCOMES:
Symptoms of post-traumatic Stress Disorder per PSS-SR (questionnaire) and CAPS (structured interview) | Four months, seven months, 14 moths, two years
Symptoms of depression as per the Beck Depression Inventory (BDI) | Four months, seven months, 14 moths, two years

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Y Shalev, M.D., Principal Investigator — Hadassah Medical Organization; Yossi Israeli - Shalev, M.A., Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization Jerusalem Israel, Jerusalem, Israel

REFERENCES:
- [Result] Shalev AY, Ankri YL, Peleg T, Israeli-Shalev Y, Freedman S. Barriers to receiving early care for PTSD: results from the Jerusalem trauma outreach and prevention study. Psychiatr Serv. 2011 Jul;62(7):765-73. doi: 10.1176/ps.62.7.pss6207_0765. PMID 21724790
- [Result] Shalev AY, Ankri Y, Israeli-Shalev Y, Peleg T, Adessky R, Freedman S. Prevention of posttraumatic stress disorder by early treatment: results from the Jerusalem Trauma Outreach And Prevention study. Arch Gen Psychiatry. 2012 Feb;69(2):166-76. doi: 10.1001/archgenpsychiatry.2011.127. Epub 2011 Oct 3. PMID 21969418
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- [Derived] van der Mei WF, Barbano AC, Ratanatharathorn A, Bryant RA, Delahanty DL, deRoon-Cassini TA, Lai BS, Lowe SR, Matsuoka YJ, Olff M, Qi W, Schnyder U, Seedat S, Kessler RC, Koenen KC, Shalev AY; International Consortium to Predict PTSD. Evaluating a screener to quantify PTSD risk using emergency care information: a proof of concept study. BMC Emerg Med. 2020 Mar 2;20(1):16. doi: 10.1186/s12873-020-00308-z. PMID 32122334
- [Derived] Shalev AY, Ankri Y, Gilad M, Israeli-Shalev Y, Adessky R, Qian M, Freedman S. Long-term outcome of early interventions to prevent posttraumatic stress disorder. J Clin Psychiatry. 2016 May;77(5):e580-7. doi: 10.4088/JCP.15m09932. PMID 27135249